CLINICAL TRIAL: NCT00053001
Title: A Phase II Study on the Effectiveness of Thalomid (Thalidomide) Combined With Procrit (Erythropoietin) for the Treatment of Anemia in Patients With Low and Intermediate Risk-1 (IPSS Score Less Than or Equal to 1.5) Myelodysplastic Syndromes
Brief Title: Thalidomide and Epoetin Alfa in Treating Anemia in Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fallon Clinic (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: FALLON-PR01-09-010; CDR0000258753 (Registry Identifier: PDQ (Physician Data Query)); CELGENE-PR01-09-010; ORTHO-PR01-09-010; FALLON-757
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-10

CONDITIONS: Anemia; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; previously treated myelodysplastic syndromes; anemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; childhood myelodysplastic syndromes
MeSH Terms: conditions — Anemia; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Epoetin Alfa; Thalidomide

INTERVENTIONS:
Biological: epoetin alfa
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop or slow the growth of cancer cells. Epoetin alfa may stimulate red blood cell production. Combining thalidomide with epoetin alfa may improve anemia, decrease the need for blood transfusions, and improve the quality of life in patients with myelodysplastic syndrome.

PURPOSE: Phase II trial to study the effectiveness of combining thalidomide with epoetin alfa in treating anemia in patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the combination of epoetin alfa and thalidomide improves the anemia and/or decreases the need for red cell transfusion in patients with low- or intermediate-risk myelodysplastic syndromes.
* Determine whether this regimen improves the bone marrow morphology and cytogenetics, alters the natural history of the disease, and reduces the frequency of leukemic transformation in these patients.
* Evaluate whether this regimen improves pathophysiologic parameters (e.g., apoptosis, tumor necrosis factor-alpha concentration, microvessel density, vascular endothelial growth factor, and cytotoxic T lymphocytes) in the bone marrow of these patients.
* Determine the safety of this regimen in these patients.

OUTLINE: Patients receive epoetin alfa subcutaneously (SC) once weekly for 8 weeks. After 8 weeks, patients unresponsive to epoetin alfa alone receive oral thalidomide once daily in addition to epoetin alfa SC once weekly for a maximum of 24 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 30-40 patients will be accrued for this study within 2 years..

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndromes

  * Newly diagnosed OR
  * Prior treatment was unsuccessful, including treatment with chemotherapy
* International prognostic scoring system score no greater than 1.5
* Hemoglobin no greater than 10 g/dL (untransfused) AND/OR
* Received at least 3 units of packed red blood cells for symptomatic anemia within the past 6 weeks

PATIENT CHARACTERISTICS:

Age

* Over 21

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 6 months

Hematopoietic

* See Disease Characteristics
* No prior bleeding disorder

Hepatic

* Bilirubin less than 2 mg/dL
* ALT/AST less than 2 times upper limit of normal

Renal

* Creatinine less than 1.5 mg/dL

Cardiovascular

* No prior clinically significant heart disease
* No uncontrolled hypertension
* No recent thromboembolic disease (e.g., deep vein thrombosis)

  * Prior thromboembolic events allowed provided event occurred at least 6 weeks prior to study and patient is on anticoagulants and is clinically stable

Pulmonary

* No unstable pulmonary disease
* No recent pulmonary embolism
* No active pulmonary infection

Neurologic

* No pre-existing peripheral neuropathy greater than grade 2
* No sustained neurologic deficit
* No epilepsy

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods (including 1 highly effective method) of contraception for at least 4 weeks before, during, and for at least 4 weeks after study completion
* No active infection
* No concurrent illness that would obscure toxicity or dangerously alter drug metabolism
* No other serious concurrent medical illness
* No uncontrolled diabetes mellitus
* No other malignant disease (except non-melanoma skin cancer or carcinoma in situ of the cervix) unless in complete remission and off therapy for that disease for more than 1 year
* No known hypersensitivity to mammalian cell-derived products or human albumin

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 4-6 weeks since prior therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Leb, MD, Study Chair — Fallon Clinic
Locations (2):
- United States (2):
  - Fallon Clinic at Worcester Medical Center, Worcester, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts